CLINICAL TRIAL: NCT00344890
Title: A Safety and Efficacy Comparison of Preservon Treated Allograft Bone Dowels Versus Traditional Freeze-Dried Allograft Bone Dowels for Fusion of Degenerated Cervical Intervertebral Discs in the Treatment of Cervical Radiculopathy or Myelopathy
Brief Title: Safety Study of Preservon-Treated Bone Implants for Cervical Fusion in the Treatment of Cervical Radiculopathy or Myelopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR06-001; WIRB Protocol #20061453
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Radiculopathy; Myelopathy
Keywords: Cervical fusion; Anterior Cervical Discectomy and Fusion; ACDF
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases; Klippel-Feil Syndrome | interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preservon (Experimental)
  Interventions: Procedure: Anterior Cervical Discectomy and Fusion
- Control (Active Comparator)
  Interventions: Procedure: Anterior Cervical Discectomy and Fusion

INTERVENTIONS:
Procedure: Anterior Cervical Discectomy and Fusion — 1,2,3,or 4 level surgery

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Preservon(TM) treated allograft bone dowels to traditional freeze-dried allograft bone dowels (control) for fusion of degenerated cervical intervertebral discs in the treatment of cervical radiculopathy or myelopathy.

Patient follow-up will be conducted at 6 weeks, 3 months, and 6 months. At 3 months after surgery, the implanted bone dowels will be assessed for subsidence; at 6 months after surgery, the implanted bone dowels will be assessed for fusion. Patients will complete questionnaires and x-rays taken at each visit.

The degree of subsidence and rate of fusion will be assessed based on the evaluation of the x-rays taken. The x-ray evaluation will be conducted by a neurosurgeon who is blinded to the type of treatment that each patient has received.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature
* Patient has confirmed radiculopathy or myelopathy
* Pain unresponsive to non-operative treatment
* Radicular pain in either or both upper extremities
* Neurological deficit in distribution of nerve root from C3/4 to C6/7
* Patient's lateral cervical spine x-rays show inferior aspect of lowest vertebral body to be fused
* Patient agrees to comply with protocol
* Patient can provide voluntary informed consent and follow-up information

Exclusion Criteria:

* Patient has previous cervical spine surgery
* Patient requires concurrent posterior surgery at level to be treated, or anterior and posterior surgery at any other cervical level
* Patient has clinically compromised vertebral body structure
* Patient has multi-level fixed/ankylosed cervical spine
* Patient has signs of significant instability at level to be treated or adjacent level
* Patient has history of metabolic bone disease
* Patient is taking chronic oral/IV corticosteroid therapy OR medications that potentially interfere with bone/soft tissue healing
* Patient has progressive neuromuscular disease, rheumatoid arthritis, active malignancy, OR any other condition that interferes with self-assessment of pain, function, or quality of life
* Patient has OPLL at any level
* Patient has active infection, local or systemic
* Patient is pregnant or considering pregnancy (x-ray requirements)
* Patient is participating in another investigational study
* Patient belongs to vulnerable population

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-09; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Degree of subsidence | 3 months post-op
Rate of fusion | 6 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E. Mathern, M.D., Principal Investigator — VCU Medical Center
Locations (1):
- VCU Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Graham RS, Samsell BJ, Proffer A, Moore MA, Vega RA, Stary JM, Mathern B. Evaluation of glycerol-preserved bone allografts in cervical spine fusion: a prospective, randomized controlled trial. J Neurosurg Spine. 2015 Jan;22(1):1-10. doi: 10.3171/2014.9.SPINE131005. PMID 25360528